CLINICAL TRIAL: NCT04042142
Title: In-depth Studies of Glucagon Resistance on Hepatic Glucose, Fatty Acid and Triglyceride Kinetics and Generation of Toxic Lipid Intermediates in NAFLD and NASH.
Brief Title: Glucagon Resistance in Patients With NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Council for Independent Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 230279
Record Dates: First submitted 2019-05-23; First posted 2019-08-01 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2020-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis; Glucose Metabolism Disorders
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Glucose Metabolism Disorders | interventions — Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy overweight subjects (Active Comparator): MR spectroscopy verified no steatosis
  Interventions: Other: glucagon
- Subjects with non-alcoholic fatty liver disease (Active Comparator): MR spectroscopy verified steatosis, no steatohepatitis on liver biopsy
  Interventions: Other: glucagon
- Subjects with non-alcoholic steatohepatitis (Active Comparator): MR spectroscopy verified steatosis, steatohepatitis on liver biopsy
  Interventions: Other: glucagon

INTERVENTIONS:
Other: glucagon — Infusion of low dose glucagon and high dose glucagon during simultaneous somatostatin infusion and replacement doses of insulin and growth hormone. Infusion of palmitate, VLDL-triglyceride and glucose tracers.

SUMMARY:
The investigators propose that the sensitivity to glucagon in hepatic lipid metabolism is impaired in subjects with non-alcoholic fatty liver disease (NAFLD) and steatohepatitis (NASH). Moreover, they propose a dys-coordinated, reduced glucagon sensitivity in hepatic lipid metabolism and endogen glucose production in patients with NAFLD and NASH compared with healthy subjects and patients with simple steatosis. This reduced sensitivity may be the basis of a more severe dyslipidemia and the production of increased concentrations of toxic lipid intermediates in plasma and muscle tissue. The study will include healthy subjects with obesity and subjects with simple steatosis and NASH, tested at basal glucagonemia and moderate hyperglucagonemia to mimic insulin resistant levels during simultaneous somatostatin infusion and replacement doses of insulin and growth hormone. Infusion of palmitate, VLDL-triglyceride and glucose tracers in combination with indirect calorimetry as well as skeletal and adipose tissue biopsies will be employed to assess free fatty acid and VLDL-triglyceride kinetics (turnover, and oxidation) and hepatic fatty acid-esterification.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 28 kg/m2
* steatosis FF% > 5,6% on MR spectroscopy for NAFLD and NASH groups

Exclusion Criteria:

* active smoking
* pregnancy
* comorbidity other than hypertension and hyperlipidemia
* participation in other radioactive isotope studies within the past 3-5 months (depending on radiation dose)
* blood donation (within 3 months)

Ages: 38 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
VLDL-triglyceride kinetics (appearance rate (µmol/min) and oxidation (µmol/min)) | 30 minutes at steady-state
  Ex vivo labeled VLDL [14C]-triolein tracer technique. Oxidation is measured by specific activity in exhaled air.
Endogen glucose production (mmol/kg/min) | 30 minutes at steady-state
  3-3H glucose tracer technique

SECONDARY OUTCOMES:
LPL-activity (lipoprotein lipase, µmol/h) | 30 minutes at steady-state
  Measured by the 'glycerol-stabilized substrate' method
VLDL-triglyceride-fatty acid uptake in muscle and fatty tissue (%) | 30 minutes at steady-state
  Measurement of fatty acid concentration and specific activity in muscle- and adipose tissue biopsies
Expression of relevant genes in tissues | 30 minutes at steady-state
  PCR in muscle- and adipose tissue biopsies
Fatty acid turnover (µmol/min) | 30 minutesat steady-state
  Infusion af [9,10-3H] palmitate and measurement of specific activity in muscle and adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Sara Heebøll, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Danmark, Denmark

REFERENCES:
- [Derived] Heeboll S, Wegener G, Gronbaek H, Nielsen S. Comparable glucagon-stimulated amino acid suppression in individuals with and without hepatic steatosis or steatohepatitis. Am J Physiol Endocrinol Metab. 2024 Dec 1;327(6):E679-E685. doi: 10.1152/ajpendo.00187.2024. Epub 2024 Sep 18. PMID 39291967
- [Derived] Heeboll S, Risikesan J, Ringgaard S, Kumarathas I, Sandahl TD, Gronbaek H, Sondergaard E, Nielsen S. Impaired Glucagon-Mediated Suppression of VLDL-Triglyceride Secretion in Individuals With Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD). Diabetes. 2022 Nov 1;71(11):2402-2411. doi: 10.2337/db22-0313. PMID 36001750